CLINICAL TRIAL: NCT03310112
Title: Mindfulness Training in U.S. Army Cohorts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Amishi Jha, Associate Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20170243
Record Dates: First submitted 2017-10-03; First posted 2017-10-16 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Psychological Stress; Anxiety; Post Traumatic Stress Disorder; Depression; Cognitive Change
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into three groups: (i) a 4-week MT group (MT4, n = 40) that will receive MBAT in 4, 2-hour sessions over 4 weeks; (ii) a 2-week MT group (MT2, n = 40) that will receive MBAT in 4, 2-hour sessions over 2 weeks; (iii) a no-training control group that will be tested before and after a no-training interval (NTC4, n = 40). After the end of the course sessions, participants from the training groups will still be assigned homework exercises until third testing session (T3). Hence, the MBAT program consists of delivery of the MBAT course, including homework mindfulness practice, and followed by an interval of homework mindfulness practice without course meetings.
  The design relies on group randomization at the level of individual military cohort units. This is due to the military requirement that organic unit structure can be maintained during testing and course session scheduling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4-week MBAT (Experimental): Participants will engage in Mindfulness-Based Attention Training (MBAT) in 4, 2-hour training classes over 4 weeks.
  Interventions: Behavioral: 4-week MBAT
- 2-week MBAT (Active Comparator): Participants will engage in Mindfulness-Based Attention Training (MBAT) in 4, 2-hour training classes over 2 weeks.
  Interventions: Behavioral: 2-week MBAT
- No training control (NTC) (No Intervention): Participants will receive no intervention but will be tested before and after a no-training interval.

INTERVENTIONS:
Behavioral: 4-week MBAT — The training is known as Mindfulness-Based Attention Training, or MBAT. The MBAT program is based on the principles of Mindfulness-Based Stress Reduction, but contextualized for military personnel using themes relevant to military life. The training content is comprised of four central themes: concentration, body awareness, open monitoring, and compassion. This content will be delivered in 4, 2-hour sessions over 4 weeks. Participants will be assigned homework mindfulness practice during the interval of course delivery as well as for the few weeks following the end of the course.
  Arms: 4-week MBAT
Behavioral: 2-week MBAT — The training is known as Mindfulness-Based Attention Training, or MBAT. The MBAT program is based on the principles of Mindfulness-Based Stress Reduction, but contextualized for military personnel using themes relevant to military life. The training content is comprised of four central themes: concentration, body awareness, open monitoring, and compassion. This content will be delivered in 4, 2-hour sessions over 2 weeks. Participants will be assigned homework mindfulness practice during the interval of course delivery as well as for the few weeks following the end of the course.
  Arms: 2-week MBAT

SUMMARY:
This project aims to contextualize delivery of mindfulness training to U.S. Army personnel, evaluate its effectiveness on measures of executive functions and psychological well-being, and determine best practices for its delivery.

DETAILED DESCRIPTION:
Background: An individual's success in the U.S. Army relies on many factors including the integrity of executive functions (EFs). EFs comprise a complex, multi-faceted brain system necessary to pay attention, overcome habitual and automatic behaviors, regulate mood, and ensure that current behavior is in line with short and long-term goals.Yet, protracted periods of high uncertainty, high demands, and high stress can lead to decreases in the efficiency and availability of EFs. Given the high demands and psychological vulnerabilities that U.S. Army personnel may face, it is critical to provide them with training programs to protect against degradation of EFs (particularly attention and working memory) over high-stress, high-demand intervals. Prior research on mindfulness training (MT) in civilians and military servicemembers showed that MT can effectively protect against degradation in attention and working memory and benefit psychological well-being over high-demand intervals.

Problem: While being successful, prior MT programs required a considerable amount of time dedicated to training (e.g., 24-hour training) and it is challenging to integrate these long programs into the busy schedule of the U.S. Army personnel. To accommodate the time constraints, the principal investigator together with a mindfulness expert developed a short-form mindfulness training program contextualized for the U.S. Army; the program consists of 8-hour training and is known as MBAT, Mindfulness-Based Attention Training.

Project Goal: The present study aims to investigate the best practices for delivery of a short-form mindfulness training to U.S. Army Cohorts. Specifically, the present study will examine the best delivery structure for the MBAT by comparing MBAT course delivered in 2 weeks vs. 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* U.S. Army personnel
* Able to understand and provide signed informed consent

Exclusion Criteria

* Non-controlled sever medical disease that might interfere with the performance in the study
* Any other condition that the investigator might deem problematic for the inclusion of the volunteer in a training study of this nature

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Change in Sustained Attention to Response Task (SART) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  The SART is used to assess attentional performance and mind wandering (i.e., off-task thinking which is typically self-generated and compromises the performance of the task at hand). The task uses a continuous performance paradigm involving button presses to frequently presented non-targets (numbers 1, 2, 4, 5, 6, 7, 8, and 9) but requires the participants to withhold their motor response to the infrequent target (number 3). Withholding responses only to infrequent targets encourages a pre-potent response and mind wandering. Real-time subjective experience of mind wandering during SART is assessed through experience-sampling probes randomly presented throughout the task.
Change in Working Memory Task with Affective Distraction (WMDA) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  The WMDA is used to assess the ability to hold information in working memory while overcoming emotional reactivity and distraction. Specifically, participants are presented with a memory item that they need to memorize and hold in memory during a delay interval. During the delay, emotionally negative or neutral scene images are presented. The negative images are combat scenes from Iraq or Afghanistan and the neutral images are non-combat scenes.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire depression scale (PHQ) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  PHQ is used as a valid diagnostic and severity measure for depressive disorders.
Change in Generalized Anxiety Disorder assessment (GAD-7) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  GAD is used as a screening tool and severity measure for generalized anxiety disorder.
Change in PTSD Checklist_Military (PCLM) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  PCLM assesses the symptoms of Post-Traumatic Stress Disorder in military personnel.
Change in the Pittsburgh Sleep Quality Index (PSQI) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  PSQI assesses sleep quality and disturbances in seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Change in Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  AUDIT-C allows to identify people who are hazardous drinkers or have active alcohol use disorders.
Change in Brief Resilience Scale (BRS) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  BRS assesses the ability to bounce back or recover from stress.
Change in Perceived Stress Scale (PSS) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  PSS assesses the degree to which situations in one's life are viewed as stressful within the past month. Individual items assess feelings of stress, nervousness, irritation at life's hassles, and perceptions of one's own coping and control over a situation.
Change in Positive and Negative Affect Scale (PANAS) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  PANAS assesses positive and negative affect. It consists of a list of descriptors of positive (e.g., 'interested', 'enthusiastic') and negative (e.g., 'irritable', 'upset') affects. Items are rated on a 5-point scale (1 = very slightly or not at all, 5 = extremely), according to how participants feel. The Positive Affect scale reflects the extent to which a person feels enthusiastic, active, and alert; the Negative Affect scale reflects unpleasant mood states, such as anger, disgust, and fear.
Change in Adult Decision-Making Competence scale (Sunk Costs questionnaire) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  Sunk Costs assesses resistance to framing, recognizing social norms, under/overconfidence, applying decision rules, risk perception, resistance to sunk costs, and path independence. A variant of this measure assessing resistance to sunk costs in a military context may be used.
Change in Cognitive Failures Questionnaire (CFQ) | Change from the pre-intervention baseline (testing 1) to the immediate post-intervention (testing 2; either 2 weeks or 4 weeks according to the group) and the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  CFQ assesses the frequency of committing minor, everyday mistakes.
Change in Five-Facet Mindfulness Questionnaire (5FMQ) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  5FMQ assesses five major measures of mindfulness, including non-judgment of experience, non-reactivity to inner experience, observing emotions, acting with awareness, and describing feelings in words.
Change in Emotion Regulation Questionnaire (ERQ) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  ERQ assesses individual differences in two emotion regulation strategies: expressive suppression and cognitive reappraisal.
Change in Combat Experiences Scale (CES) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  CES assesses how many different experiences someone had while deployed and in combat.
Change in Rumination and Response Scale (RRS) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  RRS assesses two aspects of rumination: brooding and reflective pondering
Change in Self-Compassion Questionnaire (SCQ) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  SCQ assesses various facets of self-compassion
Change in Mind Wandering Questionnaire (MWQ) | Change from the pre-intervention baseline (testing 1) to the long-term post-intervention (testing 3), which is an average of 8 weeks from the baseline.
  MWQ assesses common experiences related to distraction and mind-wandering.
Practice logs | Participants will complete paper practice logs tracking their daily practice (i.e., minutes) from the beginning of the MBAT through study completion (testing 3), which is an average of 8 weeks after beginning of the intervention.
  Practice logs will be used to keep track of participants daily mindfulness practice.
Motivation | Participants answer the motivation questions during the long-term post-intervention (testing 3) testing session, which is an average of 8 weeks from the baseline.
  Five questions regarding motivation to complete the testing session

CONTACTS AND LOCATIONS:
Overall Officials: Amishi P Jha, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jha AP, Morrison AB, Dainer-Best J, Parker S, Rostrup N, Stanley EA. Minds "at attention": mindfulness training curbs attentional lapses in military cohorts. PLoS One. 2015 Feb 11;10(2):e0116889. doi: 10.1371/journal.pone.0116889. eCollection 2015. PMID 25671579
- [Background] Jha, AP, Morrison, AB, Parker, SC, & Stanley, EA. Practice is protective: Mindfulness training promotes cognitive resilience in high-stress cohorts. Mindfulness. 2016; 7(1), 1-13. doi: 10.1007/s12671-015-0465-9.
- [Background] Jha AP, Krompinger J, Baime MJ. Mindfulness training modifies subsystems of attention. Cogn Affect Behav Neurosci. 2007 Jun;7(2):109-19. doi: 10.3758/cabn.7.2.109. PMID 17672382
- [Background] Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. Emotion. 2010 Feb;10(1):54-64. doi: 10.1037/a0018438. PMID 20141302
- [Background] van Vugt MK, Jha AP. Investigating the impact of mindfulness meditation training on working memory: a mathematical modeling approach. Cogn Affect Behav Neurosci. 2011 Sep;11(3):344-53. doi: 10.3758/s13415-011-0048-8. PMID 21732031
- [Derived] Zanesco AP, Denkova E, Rogers SL, MacNulty WK, Jha AP. Mindfulness training as cognitive training in high-demand cohorts: An initial study in elite military servicemembers. Prog Brain Res. 2019;244:323-354. doi: 10.1016/bs.pbr.2018.10.001. Epub 2018 Nov 27. PMID 30732844